CLINICAL TRIAL: NCT01276145
Title: Prevalence Of Internal Pudendal Artery Disease In Patients With Erectile Dysfunction Undergoing Diagnostic Coronary Angiography
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-292-A
Record Dates: First submitted 2011-01-10; First posted 2011-01-13 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: To Assess the Presence of Internal Pudendal Artery Disease in Patients With Erectile Dysfunction Undergoing Coronary Angiography
Keywords: pudendal artery disease; erectile dysfunction; coronary angiography; coronary disease; cardiac
MeSH Terms: conditions — Erectile Dysfunction; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Subjects in this study have recently had or are scheduled for a coronary angiography as part of their normal, routine medical care. This procedure uses x-ray imaging to see the inside of the heart's blood vessels.

This research study will evaluate the possible relationship between erectile dysfunction and vascular disease (diseases of the veins). In order to look at this possible relationship, subjects will complete a questionnaire which will ask questions regarding their sexual activity. Additionally, we will gather information from their medical records and take extra images during the coronary angiography procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age >40 years

Exclusion Criteria:

1. Creatinine Clearance < 60mL/min/1.73m2
2. Age>85
3. History of penile prosthesis
4. History or pelvic radiation or trauma

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only stable patients scheduled to undergo clinically indicated coronary angiography under non-emergent conditions will be approached for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
To assess the presence of internal pudendal artery disease in patients with erectile dysfunction undergoing coronary angiography | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Atman Shah, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States